CLINICAL TRIAL: NCT02200796
Title: Role of Dietary Protein in a Familiar Breakfast Meal on Subjective Satiety, Food Intake and Thermic Effect of Food in Normal Weight and Overweight/Obese Children
Brief Title: Role of Dietary Protein on Satiety, Food Intake and Thermic Effect of Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Assistant Professor and Director, Food Intake Regulation & Satiety, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: tempID
Record Dates: First submitted 2014-07-20; First posted 2014-07-25 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Overweight; Obesity
Keywords: Dietary Protein; Satiety; Food Intake; Thermic Effect of Food; Diet Induced Thermogenesis
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Protein Meal (Experimental): Low Protein Test Meal (15 g)
  Interventions: Other: Low Protein Meal
- Moderate Protein Meal (Experimental): Moderate Protein Meal (30 g)
  Interventions: Other: Moderate Protein Meal
- High Protein Meal (Experimental): High Protein Meal (45g)
  Interventions: Other: High Protein Meal
- Control Meal (Experimental): High Carbohydrate Control Meal (7 g of protein)
  Interventions: Other: Control Meal

INTERVENTIONS:
Other: Control Meal — High carbohydrate meal
  Arms: Control Meal
Other: Low Protein Meal — Omelet with 15 g of protein
  Arms: Low Protein Meal
Other: Moderate Protein Meal — Omelet with 30 g of protein
  Arms: Moderate Protein Meal
Other: High Protein Meal — Omelet with 45 g of protein
  Arms: High Protein Meal

SUMMARY:
Objectives: To determine the effect of protein content of familiar breakfast meals on subjective appetite, food intake (FI), glycemic response and Thermic Effect of Food (TEF) in normal weight (NW) and overweight (OW)/obese (OB) children.

Specific Objectives:

1a.To determine the effect of familiar breakfast meals (450 kcal containing eggs and varying in protein content (15, 30, and 45g) on subjective appetite, glycemic response and food intake at a test meal 4 h later in NW and. OW/OB children.

1b. To describe the effect of isocaloric (450 kcal) familiar breakfasts either high in protein (optimal protein from Objective 1a) or low in protein on TEF and substrate utilization over 5 h in NW and OW/OB children.

DETAILED DESCRIPTION:
Hypothesis: The investigators hypothesize that increasing the high-quality protein content of a breakfast meal will dose dependently increase subjective satiety, lower FI and glycemic response, and increase the TEF in both NW and OW/OB children.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between the ages of 9 and 14 y
* Only peri-pubertal girls
* Normal body weight (between the 5th and 85th BMI percentile for age and gender)
* OW/OB (>85th BMI percentile for age and gender)

Exclusion Criteria:

* Food sensitivities
* Food allergies
* Dietary restrictions
* Health, learning, emotional or behavioural problems
* On any medication

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
1a) Ad libitum food intake (in kcal) | Four hours after breakfast

SECONDARY OUTCOMES:
1b) The thermic effect of a high versus low protein meal | Resting energy expenditure (REE) at baseline and up to five hours post test meal
  REE will be determined by indirect calorimetry under a ventilated hood (ParvoMedics TrueOne 2400 automated metabolic gas analysis system, Parvo Medics, USA)
Subjective Appetite | Assessed every 15 min for 4 h
Blood glucose response | Measures at 15, or 60 min intervals for 4 h
  Finger prick capillary blood glucose (in mmol/L) at baseline, after breakfast (30 min), at 60 min, and in 1h intervals onward

CONTACTS AND LOCATIONS:
Locations (1):
- Ryerson University, FIRST Labaratory. 350 Victoria Street, Toronto, Ontario, Canada